CLINICAL TRIAL: NCT01026025
Title: A Prospective, Multi-Center Evaluation of Endo GIA Staplers With Endo GIA Single Use Loading Units (SULUs) With Duet TRS TM in a Pulmonary Resection
Brief Title: Duet TRS Used in Pulmonary Resections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor is no longer pursuing this study
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Stephanie Marcucio, Senior Clinical Research Associate, Covidien
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS09003
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: lobectomy; segmentectomy; pulmonary resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duet TRS (Experimental): This is a single arm study.
  Interventions: Device: Duet TRS

INTERVENTIONS:
Device: Duet TRS — This is a single arm study.

SUMMARY:
The objectives of this clinical trial are to estimate the incidence and duration of air leaks and the incidence of prolonged air leaks (defined as > 5 days by the Society for Thoracic Surgery) when using the ENDO GIA Staplers with ENDO GIA Single Use Loading Units (SULUs) buttressed with Duet TRS TM in an anatomic pulmonary resection via Video Assisted Thoracoscopic Surgery (VATS). Anatomic pulmonary resection is defined as either a lobectomy or segmental resection. Results of the study will be compared to contemporary literature for a similar population.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older
* The patient must be scheduled to undergo segmentectomy or lobectomy via Video Assisted Thoracoscopic Surgery (VATS) for a lung nodule suspicious for or clinically proven to be primary lung cancer
* The patient must be able to tolerate general anesthesia and have cardiopulmonary reserve to tolerate the procedure
* The patient must be willing and able to comply with all study requirements and have understood and signed the informed consent.

Exclusion Criteria:

* The patient is pregnant or breastfeeding
* The patient is scheduled to undergo sleeve lobectomy, wedge resection, bi-lobectomy, pneumonectomy or Lung Volume Reduction Surgery (LVRS), or lung biopsy for suspected interstitial lung disease
* The patient has received pre-operative chemotherapy or radiation therapy for the lung cancer that will be resected
* The patient is scheduled to receive intra-operative brachytherapy
* The patient has other severe illnesses that would preclude surgery such as unstable angina or myocardial infarction within 3 months
* Re-operative surgery is excluded if it is on the same side as the previous surgery
* The patient requires chest wall reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary objectives of this clinical trial are to estimate the incidence and duration of air leaks and the incidence of prolonged air leaks (defined as > 5 days)in an anatomic pulmonary resection. | intra-operative and 1 month follow up

SECONDARY OUTCOMES:
The secondary objectives are length of hospital stay, duration of chest tube following surgery and need for Heimlich valve at discharge. | discharge and 1 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Hiran C Fernando, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts